CLINICAL TRIAL: NCT06858514
Title: Adnan Menderes Unıversity
Brief Title: The Effect of Virtual Reality and Escape Rooms in Subcutaneous Injection Teaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nihal Taskiran, Aydin Adnan Menderes University, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-2003
Record Dates: First submitted 2025-03-04; First posted 2025-03-05 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality Simulation; Escape Room Games and Role Playing Gamification; Nursing Students; Subcutaneous Injection; Skill Performance; Self-Confidence
Keywords: virtual reality; Escape room; Subcutaneous ınjection

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality group (Experimental): * 24 hours after the theoretical lecture, a demonstration will be given to the students in the laboratory environment by the researcher under the supervision of the advisor,
  * All students will be allowed to practice on low-realistic models (task trainer) under the supervision of the instructor,
  * After the laboratory practice, the "Student Information Form" and "Subcutaneous Injection Knowledge Test" will be applied to the students,
  * Students will be provided with Oculus 2 Interactive Virtual Reality Goggles to play the virtual reality gamification before clinical practice (within 7 days).
  * After completing the game, the student will be asked to fill out the "Playful Experience Scale for Gamification" and "Subcutaneous Injection Knowledge Test",
  Interventions: Other: Virtual reality
- Escape room (Experimental): 24 hours after the theoretical lecture, a demonstration will be given to the students in the laboratory environment by the researcher under the supervision of the advisor,
  * All students will be allowed to practice on low-realistic models (task trainer) under the supervision of the instructor,
  * After the laboratory application, "Student Information Form" and "Subcutaneous Injection Knowledge Test" will be applied to the students,
  * Before entering the rooms, students will be informed about the "Escape Room Game Rules" by distributing forms on which the relevant articles are written,
  * After explaining the rules of the game to the students and answering their questions, the students will be randomly divided into three groups with six people in each group,
  * Each group will be given a name of its own choosing,
  * Each group will be placed in 3 separate simulation rooms (to prevent groups from being affected by each other)
  * Students will first try to complete their assigned activity
  Interventions: Other: Escape room
- Control group (No Intervention): * 24 hours after the theoretical lecture, a demonstration of the application in the laboratory environment will be carried out by the researcher under the supervision of the advisor,
  * It will be ensured that all students will perform the application on low-real models (task trainer) under the supervision of the instructor.
  * "Student Information Form" and "Subcutaneous Injection Knowledge Test" will be applied to the students All students (all groups) will perform the first subcutaneous injection in the clinical setting under the supervision of the course instructor before proceeding to the evaluation phase. This stage is an application carried out in line with the scope of the course and thus the risk of patient harm during the evaluation phase will be reduced.

INTERVENTIONS:
Other: Virtual reality — Students will watch a video about subcutaneous injection or students will play a about subcutaneous injection by virtual reality glasses.
  Arms: virtual reality group
Other: Escape room — Students will perform crossword puzzles, word hunt and matching activities related to subcutaneous injection practice.
  Arms: Escape room

SUMMARY:
Objective: This study was planned to determine the effect of gamification-based virtual reality and escape room teaching methods on nursing students' skill learning and self-confidence levels in subcutaneous injection skill training.

Type of Research: Randomized controlled experimental research Sample of the Study: The sample of the study will consist of 54 first-year nursing students enrolled in the Fundamentals of Nursing course at Aydın Adnan Menderes University Faculty of Nursing in the spring semester of the 2025-2026 academic year.

Place and Time of the Study: The study is planned to be conducted at Aydın Adnan Menderes University Faculty of Nursing between March 03, 2025 and January 31, 2026.

Materials and Method: "Student Information Form", 'SC Injection Skill Checklist', 'Subcutaneous Injection Knowledge Test', 'Self-Confidence Scale' and 'Playful Experience Scale for Gamification' will be used to collect the data. The students forming the sample will be randomized into 3 groups, 2 experimental and 1 control group, with 18 students in each group. First, the subject of subcutaneous injection application will be explained theoretically to all students for 90 minutes. After the completion of the theoretical explanation, the students in Experimental Group 1 will be taught the skill of subcutaneous injection application in the laboratory environment using the Gamification-Based Virtual Reality Application + Demonstration method, the students in Experimental Group 2 will be taught the Escape Room + Demonstration method, and the students in the Control Group will be taught the subcutaneous injection application skill in the laboratory environment using only the Demonstration method. After the completion of the theoretical lecture and laboratory applications according to their group, the subcutaneous injection application skill levels of the students in all three groups will be evaluated first in the laboratory environment with the Objective Structured Clinical Examination (OSCE) and then in the clinical environment using the Subcutaneous Injection Application Skill Checklist. Students' self-confidence levels will be determined by self-report method using the Self-Confidence Scale after all clinical applications are completed. Descriptive (number, percentage, mean, standard deviation, minimum-maximum) and comparative statistics (Chi-Square Test, Mann Whitney U Test, ANOVA, Student t, Wilcoxon Test) will be used to analyze the data. A p value less than 0.05 will be accepted for statistical significance.

DETAILED DESCRIPTION:
Nursing is a profession that requires practicality, knowledge, and professional skills. Nursing education aims to equip students with skills such as critical thinking, problem-solving, decision-making, holistic and empathic caregiving, communication, and team collaboration as well as gaining competence in knowledge, skills, and attitudes. Today's students, the majority of whom are Generation Z, prefer to participate in education actively and need alternative and innovative ways to be involved in the learning process. At the same time, due to the rapid development of technology, the speed of transfer of information and changes in student expectations, traditional education methods in nursing education have had to be replaced by innovative teaching methods in accordance with the requirements of the age. For this reason, it is necessary to use innovative active learning methods that complement traditional education methods and ensure active participation of students in the education process.

Psychomotor skills teaching in the nursing education system has an important role in enabling students to analyze and apply the theoretical knowledge they have learned, establish a relationship between theory and practice, make observations, and gain a sense of confidence. Psychomotor skill teaching starts with the instructor explaining and practicing the skill to the student in the laboratory environment using the demonstration method and continues with the student reflecting the skills learned to the individual he/she cares for in clinical practice. However, studies show that laboratory practices, which constitute the first step of psychomotor skills teaching, cannot reflect the real clinical experience, so students cannot adapt to the skills they learn in their interactions with patients in the real clinical environment. However, clinical practice is the area of the education program that causes the most anxiety for nursing students. When psychomotor skills teaching is not adequate, students feel inadequate in clinical practice, experience a lack of confidence, and are more likely to make medical errors. As a matter of fact, factors such as the high number of students and the low number of instructors, the inability to give every student the opportunity to practice, time constraints, lack of appropriate laboratory environments and models, inadequacies in clinical practice conditions, and the complex structure of services provided in health care reduce the effectiveness of teaching. This situation poses a potential threat in terms of both decreasing the quality of nursing care and jeopardizing patient safety in the future. Therefore, safe education practices that allow students to gain experience by repeating and learning from their mistakes without harming the individual in this process gain great importance. In this direction, there is a tendency to make nursing skills training more effective with methods such as real clinical scenarios, role-playing, and video demonstration by utilizing information technologies as well as traditional methods in order for students to gain competence by receiving extensive training before going into clinical practice. As a result of this trend and the recent necessity of distance education, especially technology-based methods come to the fore in psychomotor skills teaching. As a matter of fact, considering the predisposition of the new generation of students to use technology and the innovations and technological developments in education in recent years, the use of technology-based methods in nursing education is becoming mandatory today.

Although there are many techniques in technology-based teaching methods, "gamification", which is an innovative teaching technique in nursing, is one of the most popular and recommended methods recently.

One of the popular games in recent years is the escape room game. Escape room games are live-action team-based games in which players explore one or more clues in the room, solve puzzles and fulfill tasks in order to achieve a specific goal within a limited time, usually by escaping from the room. The task of the participants in this game is to find different clues, solve puzzles and complete various tasks within a limited time. In escape rooms, participants are divided into groups, and together with their groupmates, they solve puzzles, complex problems, and perform various skills to escape from the room by following the clues given to them, using critical thinking and decision-making skills, and the group that escapes the room in the shortest time is considered successful. The goal is usually to leave the room or find an object. According to the research results, the game duration of escape rooms varies between 20-120 minutes, but most studies use 60 minutes. Although the team size in escape rooms varies, teams usually consist of 3-6 people. Learning objectives in escape rooms are aimed at knowledge and skills of a specific subject, general skills, and affective goals. In some escape rooms, theoretical knowledge and clinical skills can be evaluated together.

The escape room game is used to develop knowledge and skills in the education of medical fields such as pharmacology, medicine, pharmacy, physiotherapy, interdisciplinary health education and mostly nursing. Since the method allows students to learn by doing and experiencing with a student-centered approach, it is recommended to be integrated into the nursing education curriculum. When the studies conducted with nursing students are examined; it is reported that the escape room method helps students learn the subject, such games should be included more in nursing education and the game helps them in their exams . It also enables students to control their learning environment by combining teamwork, critical thinking, time management and creativity . Reed and Ferdig (2021) evaluated student perceptions in an escape room simulation with 14 students taking a surgical nursing course and reported that students' anxiety levels decreased and they had a lot of fun with the game. In a study conducted by Anguas-Gracia et al. (2021) with 126 third-year nursing students, students completed various tasks, solved puzzles and tests within 60 minutes through a case study showing the effects of stroke. As a result of the study, they stated that the game helped the students to learn the subject, to remember the information and practices related to the subject, that they enjoyed the game, that they were motivated, and that there should be more such games in nursing. In our country, studies using escape room games in nursing education are quite limited. In a thesis study conducted with 72 nursing students in Turkey in 2023 on parenteral drug administration, patient scenarios were prepared and an escape room game was played using materials such as jigsaw puzzles, question cards, crossword puzzles and matching activities. As a result of the research, it was stated that the escape room game increased the knowledge level and skill score averages of nursing students, and the students who participated in the escape room game had positive statements about the game. As a result of the study conducted on first-year nursing students in 2024, it was determined that the escape room game increased students' patient safety knowledge levels and improved cooperation. Escape room game is a new method in nursing education and it is recommended to conduct more research showing its effect on nursing knowledge and skills.

Another method among the technologically based methods that have been widely used in recent years is gamification-based virtual reality application. This application is a simulation method in which the skill is transferred to the computer and gamified in an environment similar to real environments that make us feel like being anywhere and provide various information to our sensory organs for this. Studies have shown that gamification-based virtual reality applications increase students' motivation.This study was planned to determine the effect of gamification-based virtual reality and escape room teaching methods on nursing students' skill learning and self-confidence levels in subcutaneous injection skill training.

Hypotheses H0 (a): Gamification-based virtual reality application has no effect on students' level of learning subcutaneous injection skill.

H1 (a): Gamification-based virtual reality application has an effect on students' level of learning subcutaneous injection skill.

H0 (b): Escape room teaching technique has no effect on students' learning level of subcutaneous injection skill.

H1 (b): Escape room teaching technique has an effect on students' level of learning subcutaneous injection skill.

H0 (c): Gamification-based virtual reality application has no effect on students' self-confidence level.

H1 (c): Gamification-based virtual reality application has an effect on students' self-confidence level.

H0 (d): Escape room teaching method has no effect on students' self-confidence level.

H1 (d): Escape room teaching technique has an effect on students' self-confidence level.

ELIGIBILITY:
Inclusion Criteria:

* not graduated from health vocational high school.
* had no previous training in SC injection administration.
* no clinical experience.
* Participated in all theoretical and laboratory courses and all stages of the research on the dates when the SC injection subject was taught.
* To be a student of nursing department.
* who volunteer to participate in the research

Exclusion Criteria:

* students not participating in the evaluation phase.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Skill Evaluation | Once, 15 days after the theoretical lecture and laboratory practice.
  In the first stage, after the first clinical practice of the skills training, the subcutaneous skills learning levels of all students will be evaluated on the model in the laboratory environment. The assessment will be done by Objective Structured Clinical Examination (OSCE). OSCE, which is an approach used to evaluate skill performance, is a valid strategy used to assess students' readiness to perform the expected practices and skills at the desired level during clinical practice.In the second stage, all students will be evaluated in the second clinical practice one week after the completion of the theoretical skills training, laboratory practices according to their group and the first clinical practice. The second subcutaneous injection practice of the students in all three groups on patients in clinical practice will be evaluated by the researchers in accordance with the skill checklists.

SECONDARY OUTCOMES:
Confidence | once, up to 6 weeks (when the research is fınıshed)
  The confidence levels of students in all three groups will be evaluated using the " Self Confidence Scale". The scale consists of 33 items collected under two factors as internal self-confidence and external self-confidence. In the self-report and 5-point Likert-type scale, 17 items collected under the internal self-confidence factor are mostly related to individuals' self-confidence towards themselves, while the external self-confidence dimension consisting of 16 items is related to individuals' self-confidence towards their external environment and social life. The highest score that can be obtained from the scale is 165 and the lowest score is 33. A high score obtained from the scale indicates a high level of self-confidence. The total score obtained from the scale divided by the number of items determines the level of self-confidence. Accordingly, <2.5 indicates low self-confidence, 2.5-3.5 indicates medium self-confidence, and 3.5 and above indicates high self-confidenc

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Aydin, Şehzadeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available on request form the corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: end of the study
Access Criteria: The data that support the findings of this study are available on request form the corresponding author.